CLINICAL TRIAL: NCT07367451
Title: Effect of Propolis-Derived Flavonoid Extract on TLR4 Signaling and Inflammatory Cytokine Expression in Human Periodontal Ligament Stem Cells (PDLSCs): An In-Vitro Study
Brief Title: Effects of Propolis Flavonoids on TLR4 Signaling and Inflammation in Human PDLSCs In Vitro
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer of Oral Medicine, Periodontology, and Oral Diagnosis Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 12/2025
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Cytokine Expression
Keywords: TLR4; flavonoid-rich propolis; Periodontal ligament; stem cells

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated PDLSCs, and adding Flavonoid extract from propolis
  Interventions: Drug: Flavonoid extract from propolis
- Isolated PDLSCs, no material added
  Interventions: Other: no medication added

INTERVENTIONS:
Drug: Flavonoid extract from propolis — Preparation of Propolis Flavonoid Extract
  Concentrations for testing:
  5 µg/mL 10 µg/mL 20 µg/mL
  Groups: Isolated PDLSCs, and adding Flavonoid extract from propolis
Other: no medication added — No medication will be added to the second group
  Groups: Isolated PDLSCs, no material added

SUMMARY:
This in-vitro study evaluated the effects of a flavonoid-rich propolis extract on Toll-like receptor 4 (TLR4) signaling and inflammatory cytokine expression in human periodontal ligament stem cells (PDLSCs). PDLSCs were treated with propolis flavonoids under baseline conditions and following lipopolysaccharide (LPS)-induced inflammation, with untreated cells serving as controls. TLR4 gene expression was analyzed using PCR, while levels of pro-inflammatory cytokines (IL-1β, IL-6, and TNF-α) were quantified by ELISA. Cell viability and cytotoxicity at different extract concentrations were assessed using the MTT assay. The study aimed to determine the immunomodulatory and cytocompatible potential of propolis flavonoids in regulating inflammatory responses in PDLSCs.

ELIGIBILITY:
Inclusion Criteria:

* invitro study on Human Periodontal Ligament Stem Cells

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: in vitro study
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
TLR4 expression | 48 hours
  To evaluate the expression of TLR4 in PDLSCs after treatment with propolis flavonoid extract.